CLINICAL TRIAL: NCT02429024
Title: Assessment of SMS and Smartphone Interventions for OneTouch Reveal® Experiences
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LifeScan (Industry)
Collaborators: Bio-Kinetic Europe, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3132245
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; A1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects with type 1 and type 2 diabetes will be provided with the OneTouch Verio® Flex BGM system only over a period of 24 weeks.
- Intervention (Experimental): Subjects with type 1 and type 2 diabetes will be provided with the OneTouch Verio® Flex BGM and the OneTouch Reveal® Mobile APP system over a period of 24 weeks.
  Interventions: Device: OneTouch Reveal® Mobile APP; Device: OneTouch Verio® Flex BGMS

INTERVENTIONS:
Device: OneTouch Reveal® Mobile APP — Diabetes management application for use on a mobile phone.
  Arms: Intervention
Device: OneTouch Verio® Flex BGMS — Blood Glucose Monitoring System (BGMS)
  Arms: Intervention

SUMMARY:
Assessment of SMS and Smartphone Interventions for OneTouch Reveal® Experiences with patients with Type I and Type II diabetes.

DETAILED DESCRIPTION:
The primary objective is to demonstrate improved A1c in study subjects with type 1 and type 2 diabetes using the OneTouch Verio® Flex BGM and the OneTouch Reveal® Mobile APP system over a period of 24 weeks, compared to subjects using the OneTouch Verio® Flex BGM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years old (or the legal age of consent in the jurisdiction in which the study is taking place) to 70 years old, inclusive;
* Has an A1c ≥7.5 and ≤ 11.0% at screening visit;
* It is medically appropriate in the opinion of the investigator for the Subject to attempt to achieve a level of glycemic control in line with the ADA guidelines on glyceamic recommendations (<7.0% A1c, pre-prandial capillary glucose of 3.9-7.2mmol/l and peak post-prandial glucose of <10.0mmol/l);
* Diagnosed with T2DM or T1DM for ≥ 3 month prior to screening;
* Currently performing SMBG at home for diabetes management decisions and willing to test SMBG ≥ 1 per day if subject has Type 2 diabetes and is on AHA and/or non-insulin injectable (e.g. GLP-1) only, ≥ 2 per day if on basal insulin or premixed insulin; and test ≥ 3 times per day if subject has Type 2 diabetes and is on MDI or subject has Type 1 diabetes.
* Willing to send and receive SMS messages using a sponsor smartphone at 2 weekly intervals throughout the study (note: this inclusion applies to all subjects regardless of whether they are subsequently randomized to control or intervention)
* Is located in an area that can send and receive SMS messages and has access to a phone signal to use the 3G network as required
* On a stable dose of anti-hyperglycemic agents (AHA), including oral hypoglycemics (OAs), non-insulin injectables (e.g. GLP-1) or insulin therapy ≥ 2 months prior to screening; (Note: the definition of stable includes subjects who routinely self-adjust insulin based on 'in the moment' SMBG values. Stable does not include actual diabetes therapy changes (e.g. new oral medications, initiating insulin or changing insulin regimen, insulin to carb ratio changes or basal to bolus insulin progression)
* Anti-hyperglycemic agents (AHA)(OAs or GLP-1s) must be consistent with UK labeling for the subject's insulin type;
* Willingness to not use a CGM device during the study period;
* Willingness to notify the study staff if they become pregnant during the study;
* Willingness to practice an appropriate form of birth control during the study if of child bearing potential;
* Able to communicate (speak, read and write) in English, and able to understand and sign the required study documents;
* Have signed an informed consent (or regional equivalent) document indicating they understand the purpose and procedures of the study;

Exclusion Criteria:

* Is unlikely to be compliant with the currently prescribed diabetes regimen, in the opinion of the study staff;
* Currently pregnant or planning pregnancy within the duration of the study or breast feeding;
* Has unstable (rapidly progressing) retinopathy that in the opinion of the study staff may require surgical treatment (including laser photocoagulation) during the study
* Is currently on or received treatment during the past 3 months with Systemic corticosteroids or anti-psychotic drugs or prescription cannabinoid
* Is currently psychiatrically unstable in the opinion of the study staff
* Has known clinically significant and/or unstable medical conditions, in the opinion of the study staff, including: Cardiovascular disease, Hematological disease, Hepatic disease, Gastrointestinal disease, Endocrine/metabolic disorders and Neurologic disease
* Malignant neoplasm requiring treatment in the past 5 years, other than basal cell/squamous cell carcinoma of the skin
* History of major surgery within 6 months
* Has had any condition that in the opinion of the study staff that would complicate or compromise the study, or the well being of the Subject
* Subject is an employee of the investigator or clinical site;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
A1c change from baseline in subjects using the OneTouch Verio® Flex BGM and the OneTouch Reveal® Mobile APP system compared to subjects using only the OneTouch Verio® Flex (without Bluetooth) for 24 weeks. | 24 Weeks

SECONDARY OUTCOMES:
A1c ≤ 7.0% | 12 and 24 weeks
Change in A1c from baseline | 12 and 24 weeks
Quantity and percentage of glucose results within personalized glycemic ranges set by HCP at baseline. | 12 and 24 weeks
Percentage of patients that performed SMBG tests as instructed by HCP. | 24 weeks
OneTouch Reveal Mobile APP interaction and usage via APP analytics over 24wks. | 24 weeks

OTHER OUTCOMES:
Change in patient satisfaction ( DTSQ survey) | Baseline and 24 weeks
Number of SMS messages sent by the HCP | 24 weeks
Healthcare efficiency survey by the HCP | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mike Grady, Study Director — LifeScan
Locations (4):
- United Kingdom (4):
  - BioKinetic Europe Ltd, Belfast, Antrim
  - Diabetes Centre, Heartlands Hospital, Birmingham
  - NHS Lothian, Edinburgh
  - Highland Diabetes Institute, Inverness

REFERENCES:
- [Derived] Grady M, Katz LB, Cameron H, Levy BL. Diabetes App-Related Text Messages From Health Care Professionals in Conjunction With a New Wireless Glucose Meter With a Color Range Indicator Improves Glycemic Control in Patients With Type 1 and Type 2 Diabetes: Randomized Controlled Trial. JMIR Diabetes. 2017 Aug 7;2(2):e19. doi: 10.2196/diabetes.7454. PMID 30291092